CLINICAL TRIAL: NCT07171736
Title: VRAST: Virtual Reality Assisted Schema Therapy
Brief Title: Virtual Reality Assisted Schema Therapy
Acronym: VRAST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22810; 22810 (Other: UMCG)
Record Dates: First submitted 2025-09-08; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Schema Therapy; Virtual Reality; Imagination; Mental Imagery

STUDY DESIGN:
Intervention Model Description: The study will use a counterbalanced within-subjects crossover design, where all participants perform an assessment and then first perform one exercise (either VR or imagination), then do an assessment, following, the other exercise (either VR or imagination), next, another assessment and finally a qualitative interview. The order of exercises will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR exercise then imagination exercise (Experimental): Receiving the VR exercise first and the imagination exercise second
  Interventions: Behavioral: Virtual Reality chairwork exercise; Behavioral: Imagination exercise
- Imaginations exercise then VR exercise (Experimental): Receiving the imagination exercise first and the VR exercise second
  Interventions: Behavioral: Virtual Reality chairwork exercise; Behavioral: Imagination exercise

INTERVENTIONS:
Behavioral: Virtual Reality chairwork exercise — A chairwork exercise from schema therapy, executed in Virtual Reality
Behavioral: Imagination exercise — A regular schema therapy imagination exercise

SUMMARY:
Schema therapy helps people understand which emotional needs were not met during childhood, and how they can take care of those needs now. One important part of the therapy is the chairwork exercise, where people imagine talking to different parts of themselves (like the strict parent or the hurt child) using empty chairs. These exercises can be very helpful, but they can also be difficult for people who find it hard to imagine things in their mind.

Virtual Reality (VR) can make these exercises easier and more powerful. VR creates a 3D world that feels real, using special equipment like a headset. In this world, people can see and interact with virtual characters that represent different parts of themselves. This can make the therapy more concrete and easier to understand, especially for people who struggle with imagination.

In this study, we want to compare the regular imagination-based exercise with the chairwork exercise done in Virtual Reality. Everyone who joins the study will do both versions of the exercise-one with imagination and one with VR. The order will be random. Before and after each exercise, we will do a short assessment to see how people feel. At the end, we will also do a short interview to hear about their experience. The whole session will take about 1.5 hours.

We want to know if people experience the VR exercise differently than the regular imagination exercise. We also want to know if these differences depend on how well someone can imagine things in their mind.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate student
* 16 years or older
* A score of > 3 on (at least) one of the schema modes (Demanding Parent, Punitive Parent, and/or Vulnerable Child)

Exclusion Criteria:

* Insufficient command of the Dutch Language

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) questions about schema modes, negative and positive affect, self-compassion and self-esteem. | Pre-, mid-, and post-assessment (within timeframe of 1.5 hours)
  VAS questions based on the Schema Mode inventory, Positive and Negative Affect Schedule (PANAS), and items on self-compassion and self-esteem that were derived from ESM studies and previous VR studies.
VAS questions on therapeutic relationship, vividness, and immersion | Mid- and post-assessment (within timeframe of 1.5 hours)
  VAS questions based on the Working Alliance Inventory Short Form Revise (WAI-SR), the Vividness of Visual Imagery Questionnaire and the Igroup Presence Questionnaire (IPQ)

SECONDARY OUTCOMES:
Subjective experiences with both exercises | Post-assessment (within timeframe of 1.5 hours)
  Qualitative interview consisting of open-ended questions to explore experiences and compare their experiences with both exercises

OTHER OUTCOMES:
Mental Imagery Ability | Pre-assessment
  For moderation analyses, mental imagery ability will be measured using the Verbalizer-Visualizer Questionnaire (VVQ) and the Vividness of Visual Imagery Questionnaire (VVIQ)
Screening questionnaire of schema modes | Screening (before start of intervention)
  The Schema Mode Inventory will be used to assess scores on schema modes, for inclusion of participants (>3 on demanding parent, punitive parent, and/or vulnerable child).
Demographic characteristics | Pre-intervention (within timeframe of 1.5 hours)
  The following demographics will be collected: sex, age, received psychological treatment in the past (yes/no, if yes: what type of treatment?), currently receiving psychological treatment (yes/no), received schema therapy in the past (yes/no), currently receiving schema therapy (yes/no).

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Cleaned data will be shared via a repository after publication of the manuscript
Time Frame: After publication of the manuscript